CLINICAL TRIAL: NCT00959764
Title: A Randomized, Double-Blind, Multiple Dose, Placebo-Controlled, Parallel Group, 48-Week, Study of Oral Recombinant Salmon Calcitonin (rsCT) Compared to Salmon Calcitonin (sCT) Nasal Spray in Postmenopausal Osteoporotic Women
Brief Title: A Study Comparing Oral Calcitonin to Nasal Spray Calcitonin in Postmenopausal Osteoporotic Women
Acronym: ORACAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tarsa Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UGL-OR0801; 2008-003322-42 (EudraCT Number)
Record Dates: First submitted 2009-08-14; First posted 2009-08-17 (Estimated); Results first posted 2013-11-19 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-09

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Calcitonin; salmon calcitonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Oral calcitonin and placebo nasal spray (Experimental): Intervention: Oral calcitonin tablet (along with placebo intranasal spray)
  Interventions: Drug: Oral Calcitonin Tablets
- Intranasal calcitonin & oral placebo (Active Comparator): Intervention: Commercially available, active comparator, intranasal calcitonin-salmon (plus matching oral placebo tablet).
  Interventions: Drug: Intranasal Calcitonin
- Placebo: tablet & intranasal spray (Placebo Comparator): Intervention: Both oral matching placebo tablets and matching intranasal placebo spray
  Interventions: Drug: Placebo tablets and placebo intranasal spray

INTERVENTIONS:
Drug: Oral Calcitonin Tablets — Oral Calcitonin tablets along with matching placebo intranasal spray
  Other Names: rsCT tablets
  Arms: Oral calcitonin and placebo nasal spray
Drug: Intranasal Calcitonin — Intranasal Calcitonin Spray
  Other Names: Miacalcin and Miacalcic
  Arms: Intranasal calcitonin & oral placebo
Drug: Placebo tablets and placebo intranasal spray — Oral Placebo Tablets/Intranasal placebo spray
  Other Names: Matching placebos
  Arms: Placebo: tablet & intranasal spray

SUMMARY:
The purpose of this study is to compare the effectiveness and tolerability of two medications, calcitonin nasal spray and a tablet containing calcitonin, in postmenopausal women with osteoporosis. Osteoporosis is the term used to describe a large group of diseases, which are characterized by loss of bone density, which makes the bones weaker. Osteoporosis often occurs in postmenopausal women.

Calcitonin is a hormone found in the human body. Together with other substances, it regulates the concentration of calcium in the blood and inhibits the natural resorption of bone. Both medications in this study contain salmon calcitonin (sCT), because this form of calcitonin is more active than human calcitonin when used as a medicine.

The calcitonin Nasal Spray used in this study is registered and available to doctors in United States for the treatment of osteoporosis. The medication being tested in this study is an oral tablet form of salmon calcitonin.

DETAILED DESCRIPTION:
This was a randomized, double-blind, double-dummy, multiple dose, placebo-controlled, parallel group, 48- week, Phase III study. Women age 45 and over who were postmenopausal and had a diagnosis of osteoporosis were eligible for the study and were randomly allocated to one of three treatment groups; placebo tablets, oral rsCT tablets or calcitonin nasal spray. Each patient was given a treatment kit, which contained the study medication to which she had been assigned and a placebo of the treatment to which she was not assigned, or placebo nasal and oral preparations, as well as the required dietary supplements (calcium and vitamin D tablets). The study medication and supplements were self-administered at home. It was anticipated that approximately 545 patients would participate in the study.

EFFICACY: Bone Mineral Density (BMD) was recorded at Screening, Week 24, and Week 48. CTx-1 and N-telopeptide of collagen 1 (NTx-1), biochemical markers of bone resorption and total Procollagen type 1 N-terminal propeptide (P1NP),a marker of bone formation, were assessed at Week 0, Week 24, and Week 48. SAFETY: Adverse events were assessed at the clinic at Weeks 0, 12, 24, 36 and 48, and by interim phone calls at Weeks 4, 8, 16, 20, 28, 32, 40, 44, and 52. At Screening, Week 12, and Week 48, a physical examination, including nasal exam, was performed and specimens for safety laboratory analysis (clinical chemistry, hematology, and urinalysis) were collected. Sera for immunogenicity evaluations were collected at Baseline, Week 12, and Week 48.

EFFICACY: The primary comparison of interest was the percent change from baseline to 48 weeks in axial lumbar spine (L1 to L4) corrected BMD comparing the rsCT oral tablet group and the calcitonin nasal spray group. The model included the factors of the covariate (baseline BMD), treatment group, and center. The hypothesis to be tested was performed to examine the non-inferiority of the oral tablet group to the nasal spray group with respect to the percent change in axial lumbar L1-L4 spine corrected BMD. Specifically, the null hypothesis to be tested was: [Mean(oral) - Mean(placebo)] - 0.5 x [Mean(nasal) - Mean(placebo)] < 0 The alternative hypothesis was that the above expression was > 0, which implied that the oral tablet group was non-inferior to nasal spray group. The primary analysis of interest employed the modified intent-to-treat population.

SAFETY: Adverse events were summarized descriptively. Mean vital signs and clinical laboratory test results in each treatment group were compared using a one-way analysis of variance. Additionally, shift tables were prepared for each laboratory variable.

ELIGIBILITY:
Inclusion Criteria:

* Female and age 45 or over.
* Must have undergone the onset of spontaneous or surgical menopause. Spontaneous menopause is defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum Follicle Stimulating Hormone (FSH) levels >40 milli-international units (mIU)/milliliter (mL) or 6 weeks post-surgical bilateral oophorectomy with or without hysterectomy.
* Diagnosis of osteoporosis on the basis of an axial lumbar spine, femoral neck or total hip BMD which is below the mean for premenopausal women by a magnitude of at least 2.5 SD or 2.0 SD, if there is a documented history of a vertebral fragility fracture.
* Must have at least three contiguous lumbar vertebrae (L1-L4) that are evaluable by DXA for BMD that is, without fracture or significant degenerative disease, as determined by Bio-Imaging Technologies, Inc.
* No clinically significant abnormal findings in the medical history, physical exam or nasal exam.
* No clinically significant abnormal laboratory values at the screening assessment.

Exclusion Criteria:

* History of severe allergic disease.
* History of metabolic and other bone diseases, including osteogenesis imperfecta, osteomalacia, and Paget's disease.
* Vitamin D insufficiency defined as a 25 hydroxyvitamin D level <20 ng/mL.
* Use of any intravenous bisphosphonate in the past 24 months, or >2 doses of intravenous bisphosphonate ever.
* Use of oral bisphosphonate before randomization, including investigational bisphosphonates, unless: 1) less than 6 months of treatment and off for 6 months, or 2) 6 to 12 months of treatment and off for 2 years, or 3) More than 12 months of treatment and off for 5 years
* Use of denosumab, fluoride, or strontium, ever.
* Use of parathyroid hormone analogs or other bone metabolic agents within 1 year preceding randomization.
* Any condition or disease that may interfere with the ability to have a DXA scan or to evaluate a DXA scan, for example, severe osteoarthritis of the spine, spinal fusion, pedicle screws, history of vertebroplasty, or degenerative disease that results in insufficient number of evaluable lumbar vertebrae, or more than 1 lumbar vertebral fracture in L1 through L4. (More than 4 vertebral fractures in T4 through L4; Bilateral hip replacements)
* Use of anabolic steroids or androgens within 6 months preceding randomization.
* Use of Vitamin D metabolites and analogs, (e.g., calcitriol) within 3 months preceding randomization). Note: Vitamin D supplementation is not exclusionary.
* Use of estrogen or estrogen-related drugs, for example, tamoxifen, tibolone, or raloxifene within 3 months preceding randomization.
* Use of coumadin within 4 weeks preceding randomization or heparin within 1 week preceding randomization.
* Chronic systemic treatment with glucocorticoids, hormone replacement therapy, calcitonin or any other medication within the previous three months which, in the opinion of the Investigator, would interfere with the study.
* Clinically relevant abnormal history, physical findings or laboratory values at the pre-study screening assessment that could interfere with the objectives of the study or the safety of the patient.
* Presence of acute or chronic illness or history of chronic illness which, in the judgment of the Investigator, makes participation in the study medically inappropriate.
* Uncontrolled hypertension, significant gastrointestinal abnormalities, uncontrolled diabetes mellitus, significant coronary heart disease, any psychotic mental illness, chronic allergic rhinitis, asthma, uncorrected endocrine dysfunction, or significantly impaired hepatic, respiratory or renal function.
* History of drug or alcohol abuse, or intake of more than 30 units of alcohol weekly.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 565 (Actual)
Dates: Start 2009-06; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Krause, M.D., Study Director — Tarsa Therapeutics, Inc.
Locations (20):
- United States (9):
  - Rheumatology Associates of N. AL, P.C., Huntsville, Alabama
  - Northern California Institute for Bone Health, Inc., Oakland, California
  - Desert Medical Advances, Palm Desert, California
  - Bethesda Health Research Center/Bone Health Center of Bethesda, Bethesda, Maryland
  - 801 N. 30th Street, Suite 6718, Omaha, Nebraska
  - New Mexico Clinical Research & Osteoporosis, Albuquerque, New Mexico
  - Bone Mineral Research Center, Mineola, New York
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - University of Wisconsin-Geriatrics & Endocrinology/Medical Sciences Center, Madison, Wisconsin
- Diagnostic Consultative Centre, "Sveta Anna" EOOD Sofia (Rheumatology Outpatient Office), Sofia, Sofia, Bulgaria
- Synexus Hungary Ltd, Budapest, Hungary
- Synexus SCM Sp zoo, Wroclaw, Wroclaw, Poland
- Clinical Research Centres SA (Pty) Ltd, Gauteng, Pretoria, South Africa
- United Kingdom (7):
  - Synexus Thames Valley Clinical Research Centre, Reading, Berkshire
  - Synexus Midlands Clinical Research Centre, Edgbaston, Birmingham
  - Synexus Wales Clinical Research Centre, Llanishen, Cardiff
  - Synexus Lancashire Clinical Research Centre, Chorley, Chorley
  - Synexus Scotland Clinical Research Centre, Clydebank, Glasgow
  - Synexus Merseyside Clinical Research Centre, Waterloo, Liverpool
  - Synexus Manchester Clinical Research Centre, Manchester, Manchester

REFERENCES:
- [Result] Binkley N, Bolognese M, Sidorowicz-Bialynicka A, Vally T, Trout R, Miller C, Buben CE, Gilligan JP, Krause DS; Oral Calcitonin in Postmenopausal Osteoporosis (ORACAL) Investigators. A phase 3 trial of the efficacy and safety of oral recombinant calcitonin: the Oral Calcitonin in Postmenopausal Osteoporosis (ORACAL) trial. J Bone Miner Res. 2012 Aug;27(8):1821-9. doi: 10.1002/jbmr.1602. PMID 22437792

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from clinics in the USA,UK,Poland, Bulgaria, Hungary, and Republic of South Africa.
Pre-assignment Details: Unequal randomization was used for the study, with patients being assigned after inclusion/exclusion criteria were met.
Groups:
- Oral Calcitonin: Patients who only received oral calcitonin as an active treatment
- Nasal Calcitonin: Patients who only received nasal calcitonin as active treatment
- Placebo: Patients who did not receive any active treatment
Period: Overall Study
Arm/Group | Oral Calcitonin | Nasal Calcitonin | Placebo
Started | 271 | 185 | 109
Completed | 176 | 128 | 73
Not Completed | 95 | 57 | 36

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Calcitonin | Nasal Calcitonin | Placebo | Total
Number analyzed (Participants) | 271 | 185 | 109 | 565
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 115 | 77 | 39 | 231
  >=65 years | 156 | 108 | 70 | 334
Age Continuous [Mean (Standard Deviation); unit: years] | 66.5 (7.6) | 66.4 (7.0) | 66.5 (8.0) | 66.5 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 271 | 185 | 109 | 565
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 35 | 24 | 12 | 71
  Hungary | 29 | 16 | 9 | 54
  Poland | 59 | 45 | 33 | 137
  South Africa | 52 | 33 | 14 | 99
  Bulgaria | 21 | 15 | 9 | 45
  United Kingdom | 75 | 52 | 32 | 159

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Bone Mineral Density (BMD) of Axial Lumbar Spine
Description: Bone Mineral Density is measured by Dual-Energy X-ray Absorptiometry (DXA) body scans. Two scans were taken for each timepoint(baseline, week 24 and week 48) and the mean of the two values was entered. The primary outcome timepoint was 48 weeks, but if a patient did not complete the full study, then the 24 week BMD value was used as Last Observation Carried Forward. The percentage change from the baseline value, set as 0%, was recorded as the primary outcome measure.
Time Frame: 48 weeks
Population: Patients who were randomized, received treatment, and had at least one post-baseline BMD value measured at least 154 days after randomization.
Measure: Least Squares Mean (Standard Deviation); unit: Percentage increase from baseline
Groups:
- Oral Calcitonin: Patients who were provided active oral calcitonin and placebo nasal medication in a blinded fashion.
- Nasal Calcitonin: Patients who were provided active nasal calcitonin and placebo oral medication in a blinded fashion.
- Placebo: Patients who were provided nasal and oral placebo medication in a blinded fashion
Arm/Group | Oral Calcitonin | Nasal Calcitonin | Placebo
Number analyzed (Participants) | 189 | 140 | 82
Percentage increase from baseline | 1.53 (3.17) [-7.20 to 12.00] | 0.76 (2.91) [-7.49 to 9.10] | 0.47 (3.21) [-9.78 to 7.84]
Statistical Analysis 1: Comparison: Oral Calcitonin vs Nasal Calcitonin vs Placebo; The overall analysis across groups was an Analysis of Covariance where the study was powered to 80% with an assumption of a standard deviation of 2.5% and a two-sided 5% level of significance. For each treatment group, the BMD at 48 weeks was compared with the BMD at baseline and a % increase was calculated (baseline = 0%). This difference was subjected to the t-test. Two-sided P-value is less than or equal to 0.05 and was not adjusted as multiple comparisons were not done; Test type: Non-Inferiority or Equivalence — Assumed placebo-adjusted effect for both active treatment groups (% increase in BMD)was 1.56% and that the placebo adjusted effect for the rsCT tablets must be at least 0.5 times the placebo adjusted effect for the calcitonin nasal spray (active control treatment group). The null hypothesis to be tested was: [Mean(oral) - Mean(placebo)] - 0.5 x [Mean(nasal) - Mean(placebo)] < 0. Reference Pigeot, et al. 2003; p = 0.002, ANCOVA — The P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was <0.05; Mean Difference (Net) = 0.77, 95% CI 2-sided [0.08 to 1.45], Standard Deviation 2.5

2. Secondary Outcome: Change in Plasma C-terminal Telopeptide of Collagen 1 (CTx-1)
Description: Change from baseline in plasma CTx-1 at 24 and 48 weeks. CTx-1 is an accepted plasma biomarker as evidence of an effect on bone resorption and the effect of oral calcitonin was compared to that of intranasal calcitonin, both vs placebo.
Time Frame: 24 weeks
Population: Modified Intent-to-Treat Population
Measure: Least Squares Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Oral Calcitonin | Nasal Calcitonin | Placebo
Number analyzed (Participants) | 184 | 135 | 78
percentage change from baseline | -42.93 (41.99) | -24.64 (41.61) | -21.09 (62.46)
Statistical Analysis 1: Comparison: Oral Calcitonin vs Nasal Calcitonin vs Placebo; Same as for Primary Outcome; Test type: Non-Inferiority or Equivalence — Same as for Primary Outcome; p = 0.0006, ANCOVA — P-value not adjusted for multiple comparisons; a priori threshold for significance was 0.05; 95% confidence interval not calculated; Mean Difference (Net) = -21.84, Standard Deviation 41.99

3. Secondary Outcome: Change in Plasma CTx-1 From Baseline
Description: Percent change from baseline of plasma CTx-1 at end of study=48 weeks
Time Frame: 48 weeks
Population: Modified Intent-to-Treat Population
Measure: Least Squares Mean (Standard Deviation); unit: Percentage change from baseline
Arm/Group | Oral Calcitonin | Nasal Calcitonin | Placebo
Number analyzed (Participants) | 188 | 140 | 81
Percentage change from baseline | -29.92 (47.53) | -11.41 (40.24) | -11.83 (35.58)
Statistical Analysis 1: Comparison: Oral Calcitonin vs Nasal Calcitonin vs Placebo; Same as Primary Outcome; Test type: Non-Inferiority or Equivalence — Same as Primary Outcome; p = 0.0012, ANCOVA — p-value not adjusted for multiple comparisons; a priori threshold for statistical significance was set at 0.05; Mean Difference (Net) = -18.09, Standard Deviation 47.53 — oral calcitonin vs placebo

ADVERSE EVENTS:
Arm/Group | Oral Calcitonin | Nasal Calcitonin | Placebo
Serious Adverse Events (participants affected / at risk) | 20/263 | 9/182 | 9/104
Other Adverse Events (participants affected / at risk) | 44/263 | 146/182 | 83/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Calcitonin (N=263) | Nasal Calcitonin (N=182) | Placebo (N=104)
Angina Pectoris (Cardiac disorders) | 1 (1) | 1 (2) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric Ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholesystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Facial bone fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Arthroscopy (Investigations) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Ishaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Scar (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0)
Bunion operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Cataract operation (Surgical and medical procedures) | 1 (2) | 0 (0) | 0 (0)
cholecystectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Cystocele repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Skin lesion excision (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Therapeutic procedure (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Vaginal operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Calcitonin (N=263) | Nasal Calcitonin (N=182) | Placebo (N=104)
abdominal pain (Gastrointestinal disorders) | 44 (65) | 29 (51) | 15 (23)
abdominal pain upper (Gastrointestinal disorders) | 29 (39) | 18 (28) | 9 (13)
nausea (Gastrointestinal disorders) | 32 (40) | 15 (18) | 7 (11)
constipation (Gastrointestinal disorders) | 18 (20) | 12 (14) | 7 (8)
dyspepsia (Gastrointestinal disorders) | 19 (24) | 8 (8) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 17 (22) | 4 (5) | 7 (8)
Nasopharyngitis (Infections and infestations) | 16 (17) | 16 (16) | 10 (11)
Urinary tract Infection (Infections and infestations) | 15 (18) | 17 (21) | 4 (6)
Upper respiratory tract infection (Infections and infestations) | 11 (12) | 13 (13) | 8 (8)
Influenza (Infections and infestations) | 17 (17) | 5 (5) | 2 (2)
Rhinitis (Infections and infestations) | 6 (7) | 6 (12) | 6 (6)
Headache (Nervous system disorders) | 20 (25) | 11 (13) | 7 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (14) | 13 (15) | 3 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No